CLINICAL TRIAL: NCT02575482
Title: A Single-center, Double-blind, Placebo-controlled, Randomized, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SUVN-D4010 After Single Ascending Doses and Multiple Ascending Doses in Healthy Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of SUVN-D4010 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP140105HT4
Record Dates: First submitted 2015-10-05; First posted 2015-10-14 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Cognitive Disorders
Keywords: SUVN-D4010; serotonin 4 (5-HT4) receptor; first in human; safety; pharmacokinetics; tolerability; single dose; repeat dose
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single and Multiple ascending dose (Experimental): Single dose of SUVN-D4010 in healthy male subjects
  Interventions: Drug: SUVN-D4010
- Placebo (Placebo Comparator): Placebo in healthy male subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SUVN-D4010
  Arms: Single and Multiple ascending dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of SUVN-D4010 in healthy male subjects following single or multiple ascending doses.

DETAILED DESCRIPTION:
This is a single and multiple ascending dose study to assess the safety, tolerability and pharmacokinetics of SUVN-D4010 administered orally once a day to healthy male subjects. The study will be conducted under double blind conditions.

The primary objective is to evaluate the safety and tolerability of SUVN-D4010 following oral administration of single or multiple ascending doses and estimate the maximum tolerated dose of SUVN-D4010,if possible.

The secondary objectives are to evaluate the single and repeat dose plasma pharmacokinetics following oral administration of single and multiple ascending doses of SUVN-D4010 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 18 to 45 years with a BMI between 18 and 30 kg/m2, (inclusive).

Exclusion Criteria:

* Standard exclusion criterion for Phase 1 clinical trial in healthy subjects.
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs as judged by Investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
ECG | Range of Day 1-17
Physical exams | Range of Day 1-17
Vitals signs | Range of Day 1-17
CSSRS (suicidality) | Range of Day 1-17
  Columbia Suicidal Severity Rating Scale
Safety and tolerability of single or multiple doses of SUVN-D4010 in healthy male subjects | Range of Day 1-17
  Incidence of Treatment-Emergent Adverse Events, Laboratory parameters

SECONDARY OUTCOMES:
Area under the SUVN-D4010 plasma concentrationtime curve in a dosing interval (AUC0tau) | Day 1
Area under the SUVN-D4010 plasma concentrationtime curve from zero to infinity (AUC0inf) | Day 14
Maximum observed concentration (Cmax) and time of observation (tmax) | Day 1 and Day 14
Oral clearance (CL/F) | Day 1 and Day 14
Accumulation index following multiple dosing of SUVN-D4010 (AI) | Day 14
Elimination half life (t½) | Day 1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickerson, Principal Investigator — Research Physician
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

REFERENCES:
- [Derived] Nirogi R, Bhyrapuneni G, Muddana NR, Goyal VK, Pandey SK, Mohammed AR, Ravula J, Jetta S, Palacharla VRC. First-in-Human Studies to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Novel 5-HT4 Partial Agonist, SUVN-D4010, in Healthy Adult and Elderly Subjects. Clin Drug Investig. 2021 May;41(5):469-482. doi: 10.1007/s40261-021-01027-4. Epub 2021 Mar 31. PMID 33788154